CLINICAL TRIAL: NCT04391972
Title: Clinical Outcome of Extended-depth-of-focus Intraocualr Lens (SAV) Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-12-019
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Presbyopia
Keywords: depth and focus
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAV multifocal IOL (Other): Subjects who have cataract surgery with SAV multifocal IOL
  Interventions: Device: SAV

INTERVENTIONS:
Device: SAV — SAV multifocal intraocular lens is a implantable IOL which offers multifocal vision.

SUMMARY:
Clinical outcome of extended-depth-of-focus intraocular lens (SAV) implantation

DETAILED DESCRIPTION:
In this study, we are trying to evaluate the clinical outcome of extended-depth-of-focus intraocular lens (SAV).

ELIGIBILITY:
Inclusion Criteria:

1. Adult at the age of 21 or older at the time of the pre-operative examination and willing to have surgery on their 2nd eye within 7-28 days of their 1st eye
2. Age-related cataract
3. A patient with preoperative corneal astigmatism from IOL Master less than 1 diopters
4. A patient want presbyopia correction at the same time as cataract surgery
5. A patient has the visual potential of 20/25 or better in each eye after cataract removal and IOL implantation
6. Written informed consent to surgery and participation in the study

Exclusion Criteria:

1. Those with other diseases that can affect capsule stability such as pseudoexoliation syndrome, glaucoma, traumatic cataract
2. Pregnant woman and lactating woman
3. A patient with history of ocular trauma or ocular surgery (Intraocular surgery, refractive surgery, ocular surface surgery) in either eye
4. A patient with evidence of keratoconus or significant irregular astigmatism on pre-operative topography in either eye
5. If expectations for presbyopia correction are too high
6. Those who are not able to read and understand the informed consent (illiterate or foreigners)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-01-22 (Estimated); Study Completion 2021-01-22 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distant visual acuity | 3 months
  Visual acuity at distance with bare eyes
Uncorrected near visual acuity | 3 months
  Visual acuity at near with bare eyes

SECONDARY OUTCOMES:
Contrast sensitivity | 3 months
  Ability to recognize letter or figure at different contrast environment
Quality of Vision | 3 months
  Degree of various symptom associated with vision

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Young Chung, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea